CLINICAL TRIAL: NCT03897335
Title: The Effect of Aminophylline on Preventing Acute Kidney Injury in Pediatric Patients Undergoing Open Heart Surgery
Brief Title: Preventing Acute Kidney Injury (AKI) in Pediatric Patients
Acronym: AKI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Le Bonheur Children's Hospital (Other)
Responsible Party: Principal Investigator, Umar S. Boston, Professor UTHSC, Le Bonheur Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Acute Kidney Injury
Record Dates: First submitted 2019-02-20; First posted 2019-04-01 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Acute Kidney Injury
Keywords: Aminophylline
MeSH Terms: conditions — Acute Kidney Injury | interventions — Aminophylline; Saline Solution

STUDY DESIGN:
Intervention Model Description: 1 Patient randomization groups
  A) Group 1: Aminophylline pre CPB & immediately post cardiopulmonary bypass (CPB)
  B) Group 2: No aminophylline prophylaxis
Who Masked: Participant, Care Provider, Investigator
Masking Description: Cohort 1 will consist of all children undergoing open heart surgery for congenital heart defects with or without circulatory arrest, and Cohort 2 will consist of Orthotopic heart transplantation patients. All subjects will be randomized 1:1 to aminophylline or saline placebo. Cohort 1 will be randomized using block-stratification with stratification factors age (neonate vs infant) and circulatory arrest (yes vs no). Age will be categorized as neonates (0 to <28 days) and infants (28 days to <1 year).
  A total of 80 (60 in Cohort 1 and 20 in Cohort 2) participants are expected to be enrolled on this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aminophylline pre CPB & immediately post CPB (Active Comparator)
  Interventions: Drug: Aminophylline
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aminophylline — Aminophylline pre cardiopulmonary bypass and immediately post cardiopulmonary bypass. The dose will be Aminophylline 5 mg/kg/dose, max 350 mg slow infusion. The infusion rate duration will be standardized to 20 minutes. There will be no other aminophylline treatments for the first post-op five days.
  Arms: Aminophylline pre CPB & immediately post CPB
Drug: Placebo — The placebo group will not receive any aminophylline treatments for the first post-op five days
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects of peri-operative administration of Aminophylline versus Saline placebo in the preservation of renal function and the attenuation of renal injury in pediatric patients undergoing open heart surgery.

DETAILED DESCRIPTION:
Cardiac palliative/ correction surgeries in pediatric patients involve significant morbidity and mortality risks. Kidney function is frequently affected from cardiac surgery in these children. Studies identify the incidence of acute kidney injury (AKI) to be approximately 54% when defined by serum biomarkers (e.g. serum creatinine) and urine output criteria. The need for renal replacement therapy (RRT) for newborns and infants after cardiac surgery is reported as 2% to 17% in the literature. There are several reported risk factors for the development of AKI in this population. These are the complexities of the underlying heart disease and the surgical procedure, duration of cardiopulmonary bypass, functional single ventricle heart disease, circulatory arrest and low cardiac output syndrome in the post-operative period. AKI can cause worsening fluid overload compromising ventilation and lung function, predisposition to overwhelming infections and cytokine-mediated inflammatory state. The presence of AKI significantly increases the mortality that is associated with cardiac surgery in these very young patients, reported as high as 79% in the literature. There have been several reports suggesting that early intervention with AKI using renal replacement therapy (RRT) may improve patient mortality. Successful prevention strategies for AKI have not been reported for this high-risk population.

Adenosine has been demonstrated to regulate renal circulation and metabolism. It is a breakdown product of adenosine triphosphate/adenosine diphosphate (ATP/ADP) metabolism and accumulates in AKI. At baseline, the barely detectable renal parenchymal adenosine levels can increase to 10-100 times following an ischemic insult. These are typical seven trans-membrane spanning domains with a coupled G-protein at the intracellular end. Adenosine receptors are located ubiquitously in many tissues. Adenosine acts as a vasodilator in all other tissues but the renal parenchyma. The interaction of AT-II with adenosine converts adenosine to a vasoconstrictor in renal microvasculature. Adenosine acts on the A1 receptors (A1 R) in the afferent arterioles, causing reduced glomerular blood flow and glomerular filtration rate (GFR), as well as stimulating renin release from the kidney parenchyma. Adenosine plays an important role in generating the vasoconstrictive response in the renal vasculature to hypoxia and ischemia. Early interventions by blocking the actions of adenosine on A1 R may restore glomerular blood flow and recover GFR.

The study rationale is that Aminophylline and Theophylline are competitive non-selective inhibitors of adenosine. Therefore, even though aminophylline infusion (iv) has no effect on renal blood flow rate at baseline, it can ameliorate the decrease in renal blood flow rate following adenosine infusion. This property can improve renal function when the main mechanism of insult induces vasoconstriction. Both early and late administration of aminophylline protects renal function after ischemia-reperfusion injury in rats. Aminophylline has also been reported to successfully reverse newborn renal failure, prevent renal failure in perinatal asphyxia, and reverse acute kidney injury secondary to calcineurin induced nephropathy. Both theophylline and aminophylline have been used for prophylaxis of renal impairment during aorto-coronary bypass surgery in adults and the results have not been consistent for either a positive or negative effect. There have been no trials reported on the effect of aminophylline or theophylline to prevent or ameliorate acute kidney injury in children with congenital heart defects going through cardiac surgery.

Additionally, we are examining the components of serotonin biosynthesis to determine if these levels can act as markers of acute kidney injury in pediatric patients undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1

* All children undergoing open heart surgery for congenital heart defects with or without circulatory arrest
* Neonates (<28 days old) and infants (<1 years of age)
* Hypoplastic L heart syndrome or its variants.
* Coarctation with aortic arch hypoplasia.
* Interrupted aortic arch.
* TAPVR (Total anomalous pulmonary venous return)
* Patients with complex congenital heart defects

Cohort 2:

* Orthotopic heart transplantation patients.
* Patients ≤ 18 years of age
* Congenital heart defects
* Cardiomyopathy (Dilated/Hypertrophic/Restrictive/Left Ventricular Non-compaction)

Exclusion Criteria:

* Children under the age of 12 months undergoing bypass for any condition that is not categorized as congenital heart defect
* History of seizures
* History of significant tachyarrhythmia.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury state II/III by AKIN criteria | At 48 hours post-operative
  Acute kidney injury state II/III by AKIN criteria

SECONDARY OUTCOMES:
Urine output during post op | first 12 hours post op
  Urine output during post op
Urine output during post op | daily until 3 days post op
  Urine output during post op
Concentration of Delta serum cystatin C | 24 hours post CPB
  Delta serum cystatin C
Acute kidney injury stage | max point within post CPB 72 hours
  Acute kidney injury stage Pediatric modified Acute Kidney Injury Network criteria (pAKIN) AKI Stage I-<0.5mL (milliliter)/kg/hour for 8 hours AKI Stage II-<0.5mL/kg/hour for 16 hours AKI Stage III-<0.3mL/kg/hour for 24 hours OR Anuria for 16 hours
  Using serum creatinine and AKIN criteria

OTHER OUTCOMES:
Concentration of Delta urinary neutrophil gelatinase-associated lipocalin (NGAL) | at 2 hours post CPB.
  1 Delta urinary NGAL at 6 hours post cardiopulmonary (CPB) and Delta plasma NGAL at 2 hours post CPB.
Time to extubation (hours) | during hospitalization, up to 8 days
  Time to extubation (hours) number of hours post surgery
Time to chest closure (hours) | during hospitalization, up to 3 days
  Time to chest closure (hours) from start time of incision to chest closure during procedure
Time to discharge from cardiovascular intensive care unit (CVICU) (days) | during hospitalization, approximate 5 days
  Time to discharge from CVICU (days)
Duration of hospital stay (Days). | during hospitalization, approximate 8 days
  Duration of hospital stay (Days).
Dialysis requirement (yes/no) | during hospitalization, approximate 5 days
  Dialysis requirement (yes/no)
Time to return to preoperative weight. | during hospitalization, approximate 8 days
  Time to return to preoperative weight.
Inotropic score | at 7 days post operative
  Inotropic score Calculation of Inotropic score (IS) and Vasoactive inotropic score (VIS). IS(a) = dopamine dose (lg/kg/min) ? dobutamine dose (lg/kg/min) ? 100 9 epinephrine dose (lg/kg/min) VIS(b) = IS ? 10 9 milrinone dose (lg/kg/ min) ? 10,000 9 vasopressin dose (U/kg/ min) ? 100 9 norepinephrine dose (lg/kg/min) IS inotrope score, VIS vasoactive-inotropic score
Peritoneal dialysis catheter output. | during hospitalization, up to 8 days
  Peritoneal dialysis catheter output through study completion
Transfusion requirements intraoperatively and postoperatively | during hospitalization, up to 8 days
  Transfusion requirements intraoperatively and postoperatively through study completion
Inotropic score | at 5 days post operative
  Inotropic score Calculation of Inotropic score (IS) and Vasoactive inotropic score (VIS). IS(a) = dopamine dose (lg/kg/min) ? dobutamine dose (lg/kg/min) ? 100 9 epinephrine dose (lg/kg/min) VIS(b) = IS ? 10 9 milrinone dose (lg/kg/ min) ? 10,000 9 vasopressin dose (U/kg/ min) ? 100 9 norepinephrine dose (lg/kg/min) IS inotrope score, VIS vasoactive-inotropic score

CONTACTS AND LOCATIONS:
Locations (1):
- LeBonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1.KDIGO Clinical Practice Guideline for Acute Kidney Injury. Kidney Int. Suppl 2 ; 2012:1-138
- [Background] Bojan M, Gioanni S, Vouhe PR, Journois D, Pouard P. Early initiation of peritoneal dialysis in neonates and infants with acute kidney injury following cardiac surgery is associated with a significant decrease in mortality. Kidney Int. 2012 Aug;82(4):474-81. doi: 10.1038/ki.2012.172. PMID 22622499
- [Background] 11.Gouyon JB, Guignard JP. Glomerular filtration rates in neonates. In Oh w, Guignard JP, Baumgart S (Eds.): Nephrology and Fluid / Electrolyte Physiology, First edn (pp 79-96). Philadelphia: Saunders Elsevier 2008
- [Background] Linden J and Jacobson KA. Molecular biology and pharmacology of adenosine receptors. Cardiovascular Biology of Purines, 1-20 (Eds Burnstock G et al.) Dordrecht: Kluwer Academic Publishers.
- [Result] Rigden SP, Barratt TM, Dillon MJ, De Leval M, Stark J. Acute renal failure complicating cardiopulmonary bypass surgery. Arch Dis Child. 1982 Jun;57(6):425-30. doi: 10.1136/adc.57.6.425. PMID 7092306
- [Result] Sorof JM, Stromberg D, Brewer ED, Feltes TF, Fraser CD Jr. Early initiation of peritoneal dialysis after surgical repair of congenital heart disease. Pediatr Nephrol. 1999 Oct;13(8):641-5. doi: 10.1007/s004670050672. PMID 10502118
- [Result] Chan KL, Ip P, Chiu CS, Cheung YF. Peritoneal dialysis after surgery for congenital heart disease in infants and young children. Ann Thorac Surg. 2003 Nov;76(5):1443-9. doi: 10.1016/s0003-4975(03)01026-9. PMID 14602265
- [Result] Boigner H, Brannath W, Hermon M, Stoll E, Burda G, Trittenwein G, Golej J. Predictors of mortality at initiation of peritoneal dialysis in children after cardiac surgery. Ann Thorac Surg. 2004 Jan;77(1):61-5. doi: 10.1016/s0003-4975(03)01490-5. PMID 14726035
- [Result] Pedersen KR, Povlsen JV, Christensen S, Pedersen J, Hjortholm K, Larsen SH, Hjortdal VE. Risk factors for acute renal failure requiring dialysis after surgery for congenital heart disease in children. Acta Anaesthesiol Scand. 2007 Nov;51(10):1344-9. doi: 10.1111/j.1399-6576.2007.01379.x. PMID 17944638
- [Result] Pedersen KR, Hjortdal VE, Christensen S, Pedersen J, Hjortholm K, Larsen SH, Povlsen JV. Clinical outcome in children with acute renal failure treated with peritoneal dialysis after surgery for congenital heart disease. Kidney Int Suppl. 2008 Apr;(108):S81-6. doi: 10.1038/sj.ki.5002607. PMID 18379554
- [Result] Ronco C, Haapio M, House AA, Anavekar N, Bellomo R. Cardiorenal syndrome. J Am Coll Cardiol. 2008 Nov 4;52(19):1527-39. doi: 10.1016/j.jacc.2008.07.051. PMID 19007588
- [Result] Blinder JJ, Goldstein SL, Lee VV, Baycroft A, Fraser CD, Nelson D, Jefferies JL. Congenital heart surgery in infants: effects of acute kidney injury on outcomes. J Thorac Cardiovasc Surg. 2012 Feb;143(2):368-74. doi: 10.1016/j.jtcvs.2011.06.021. Epub 2011 Jul 27. PMID 21798562
- [Result] Gouyon JB, Guignard JP. Functional renal insufficiency: role of adenosine. Biol Neonate. 1988;53(4):237-42. doi: 10.1159/000242796. PMID 3046670
- [Result] Hall JE, Granger JP, Hester RL. Interactions between adenosine and angiotensin II in controlling glomerular filtration. Am J Physiol. 1985 Mar;248(3 Pt 2):F340-6. doi: 10.1152/ajprenal.1985.248.3.F340. PMID 3883810
- [Result] Hansen PB, Schnermann J. Vasoconstrictor and vasodilator effects of adenosine in the kidney. Am J Physiol Renal Physiol. 2003 Oct;285(4):F590-9. doi: 10.1152/ajprenal.00051.2003. PMID 12954591
- [Result] Rabb H. The promise of immune cell therapy for acute kidney injury. J Clin Invest. 2012 Nov;122(11):3852-4. doi: 10.1172/JCI66455. Epub 2012 Oct 24. PMID 23093787
- [Result] Fredholm BB, IJzerman AP, Jacobson KA, Klotz KN, Linden J. International Union of Pharmacology. XXV. Nomenclature and classification of adenosine receptors. Pharmacol Rev. 2001 Dec;53(4):527-52. PMID 11734617
- [Result] Pawelczyk T, Grden M, Rzepko R, Sakowicz M, Szutowicz A. Region-specific alterations of adenosine receptors expression level in kidney of diabetic rat. Am J Pathol. 2005 Aug;167(2):315-25. doi: 10.1016/S0002-9440(10)62977-X. PMID 16049319
- [Result] Navar LG, Inscho EW, Majid SA, Imig JD, Harrison-Bernard LM, Mitchell KD. Paracrine regulation of the renal microcirculation. Physiol Rev. 1996 Apr;76(2):425-536. doi: 10.1152/physrev.1996.76.2.425. PMID 8618962
- [Result] Vitzthum H, Weiss B, Bachleitner W, Kramer BK, Kurtz A. Gene expression of adenosine receptors along the nephron. Kidney Int. 2004 Apr;65(4):1180-90. doi: 10.1111/j.1523-1755.2004.00490.x. PMID 15086457
- [Result] Silldorff EP, Pallone TL. Adenosine signaling in outer medullary descending vasa recta. Am J Physiol Regul Integr Comp Physiol. 2001 Mar;280(3):R854-61. doi: 10.1152/ajpregu.2001.280.3.R854. PMID 11171666
- [Result] Nishiyama A, Inscho EW, Navar LG. Interactions of adenosine A1 and A2a receptors on renal microvascular reactivity. Am J Physiol Renal Physiol. 2001 Mar;280(3):F406-14. doi: 10.1152/ajprenal.2001.280.3.F406. PMID 11181402
- [Result] Okusa MD, Linden J, Macdonald T, Huang L. Selective A2A adenosine receptor activation reduces ischemia-reperfusion injury in rat kidney. Am J Physiol. 1999 Sep;277(3):F404-12. doi: 10.1152/ajprenal.1999.277.3.F404. PMID 10484524
- [Result] Lee HT, Emala CW. Systemic adenosine given after ischemia protects renal function via A(2a) adenosine receptor activation. Am J Kidney Dis. 2001 Sep;38(3):610-8. doi: 10.1053/ajkd.2001.26888. PMID 11532695
- [Result] Okusa MD, Linden J, Huang L, Rosin DL, Smith DF, Sullivan G. Enhanced protection from renal ischemia-reperfusion [correction of ischemia:reperfusion] injury with A(2A)-adenosine receptor activation and PDE 4 inhibition. Kidney Int. 2001 Jun;59(6):2114-25. doi: 10.1046/j.1523-1755.2001.00726.x. PMID 11380813
- [Result] Reece TB, Davis JD, Okonkwo DO, Maxey TS, Ellman PI, Li X, Linden J, Tribble CG, Kron IL, Kern JA. Adenosine A2A analogue reduces long-term neurologic injury after blunt spinal trauma. J Surg Res. 2004 Sep;121(1):130-4. doi: 10.1016/j.jss.2004.04.006. PMID 15313386
- [Result] Ross SD, Tribble CG, Linden J, Gangemi JJ, Lanpher BC, Wang AY, Kron IL. Selective adenosine-A2A activation reduces lung reperfusion injury following transplantation. J Heart Lung Transplant. 1999 Oct;18(10):994-1002. doi: 10.1016/s1053-2498(99)00066-2. PMID 10561110
- [Result] Odashima M, Bamias G, Rivera-Nieves J, Linden J, Nast CC, Moskaluk CA, Marini M, Sugawara K, Kozaiwa K, Otaka M, Watanabe S, Cominelli F. Activation of A2A adenosine receptor attenuates intestinal inflammation in animal models of inflammatory bowel disease. Gastroenterology. 2005 Jul;129(1):26-33. doi: 10.1053/j.gastro.2005.05.032. PMID 16012931
- [Result] Glover DK, Riou LM, Ruiz M, Sullivan GW, Linden J, Rieger JM, Macdonald TL, Watson DD, Beller GA. Reduction of infarct size and postischemic inflammation from ATL-146e, a highly selective adenosine A2A receptor agonist, in reperfused canine myocardium. Am J Physiol Heart Circ Physiol. 2005 Apr;288(4):H1851-8. doi: 10.1152/ajpheart.00362.2004. Epub 2004 Dec 9. PMID 15591104
- [Result] Day YJ, Huang L, Ye H, Li L, Linden J, Okusa MD. Renal ischemia-reperfusion injury and adenosine 2A receptor-mediated tissue protection: the role of CD4+ T cells and IFN-gamma. J Immunol. 2006 Mar 1;176(5):3108-14. doi: 10.4049/jimmunol.176.5.3108. PMID 16493070
- [Result] Vallon V, Muhlbauer B, Osswald H. Adenosine and kidney function. Physiol Rev. 2006 Jul;86(3):901-40. doi: 10.1152/physrev.00031.2005. PMID 16816141
- [Result] Gouyon JB, Guignard JP. Theophylline prevents the hypoxemia-induced renal hemodynamic changes in rabbits. Kidney Int. 1988 Jun;33(6):1078-83. doi: 10.1038/ki.1988.114. PMID 3404810
- [Result] Bakr AF. Prophylactic theophylline to prevent renal dysfunction in newborns exposed to perinatal asphyxia--a study in a developing country. Pediatr Nephrol. 2005 Sep;20(9):1249-52. doi: 10.1007/s00467-005-1980-z. Epub 2005 Jun 10. PMID 15947981
- [Result] Ng GY, Baker EH, Farrer KF. Aminophylline as an adjunct diuretic for neonates--a case series. Pediatr Nephrol. 2005 Feb;20(2):220-2. doi: 10.1007/s00467-004-1692-9. Epub 2004 Dec 4. PMID 15583947
- [Result] Jenik AG, Ceriani Cernadas JM, Gorenstein A, Ramirez JA, Vain N, Armadans M, Ferraris JR. A randomized, double-blind, placebo-controlled trial of the effects of prophylactic theophylline on renal function in term neonates with perinatal asphyxia. Pediatrics. 2000 Apr;105(4):E45. doi: 10.1542/peds.105.4.e45. PMID 10742366
- [Result] Bhat MA, Shah ZA, Makhdoomi MS, Mufti MH. Theophylline for renal function in term neonates with perinatal asphyxia: a randomized, placebo-controlled trial. J Pediatr. 2006 Aug;149(2):180-4. doi: 10.1016/j.jpeds.2006.03.053. PMID 16887430
- [Result] McLaughlin GE, Abitbol CL. Reversal of oliguric tacrolimus nephrotoxicity in children. Nephrol Dial Transplant. 2005 Jul;20(7):1471-5. doi: 10.1093/ndt/gfh785. Epub 2005 Apr 19. PMID 15840666
- [Result] Kramer BK, Preuner J, Ebenburger A, Kaiser M, Bergner U, Eilles C, Kammerl MC, Riegger GA, Birnbaum DE. Lack of renoprotective effect of theophylline during aortocoronary bypass surgery. Nephrol Dial Transplant. 2002 May;17(5):910-5. doi: 10.1093/ndt/17.5.910. PMID 11981083
- [Result] Mahaldar AR, Sampathkumar K, Raghuram AR, Kumar S, Ramakrishnan M, Mahaldar DA. Risk prediction of acute kidney injury in cardiac surgery and prevention using aminophylline. Indian J Nephrol. 2012 May;22(3):179-83. doi: 10.4103/0971-4065.98752. PMID 23087551
- [Result] Aki Y, Tomohiro A, Nishiyama A, Kiyomoto K, Kimura S, Abe Y. Effects of KW-3902, a selective and potent adenosine A1 receptor antagonist, on renal hemodynamics and urine formation in anesthetized dogs. Pharmacology. 1997 Oct;55(4):193-201. doi: 10.1159/000139528. PMID 9396079
- [Result] Yao K, Ina Y, Nagashima K, Ohno T, Karasawa A. Effect of the selective adenosine A1-receptor antagonist KW-3902 on lipopolysaccharide-induced reductions in urine volume and renal blood flow in anesthetized dogs. Jpn J Pharmacol. 2000 Nov;84(3):310-5. doi: 10.1254/jjp.84.310. PMID 11138732
- [Result] Givertz MM, Massie BM, Fields TK, Pearson LL, Dittrich HC; CKI-201 and CKI-202 Investigators. The effects of KW-3902, an adenosine A1-receptor antagonist,on diuresis and renal function in patients with acute decompensated heart failure and renal impairment or diuretic resistance. J Am Coll Cardiol. 2007 Oct 16;50(16):1551-60. doi: 10.1016/j.jacc.2007.07.019. Epub 2007 Oct 1. PMID 17936154
- [Result] Cotter G, Dittrich HC, Weatherley BD, Bloomfield DM, O'Connor CM, Metra M, Massie BM; Protect Steering Committee, Investigators, and Coordinators. The PROTECT pilot study: a randomized, placebo-controlled, dose-finding study of the adenosine A1 receptor antagonist rolofylline in patients with acute heart failure and renal impairment. J Card Fail. 2008 Oct;14(8):631-40. doi: 10.1016/j.cardfail.2008.08.010. Epub 2008 Sep 14. PMID 18926433
- [Result] Massie BM, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, Weatherley BD, Cleland JG, Givertz MM, Voors A, DeLucca P, Mansoor GA, Salerno CM, Bloomfield DM, Dittrich HC; PROTECT Investigators and Committees. Rolofylline, an adenosine A1-receptor antagonist, in acute heart failure. N Engl J Med. 2010 Oct 7;363(15):1419-28. doi: 10.1056/NEJMoa0912613. PMID 20925544
- [Result] Voors AA, Dittrich HC, Massie BM, DeLucca P, Mansoor GA, Metra M, Cotter G, Weatherley BD, Ponikowski P, Teerlink JR, Cleland JG, O'Connor CM, Givertz MM. Effects of the adenosine A1 receptor antagonist rolofylline on renal function in patients with acute heart failure and renal dysfunction: results from PROTECT (Placebo-Controlled Randomized Study of the Selective Adenosine A1 Receptor Antagonist Rolofylline for Patients Hospitalized with Acute Decompensated Heart Failure and Volume Overload to Assess Treatment Effect on Congestion and Renal Function). J Am Coll Cardiol. 2011 May 10;57(19):1899-907. doi: 10.1016/j.jacc.2010.11.057. PMID 21545947
- [Result] Morecroft I, Dempsie Y, Bader M, Walther DJ, Kotnik K, Loughlin L, Nilsen M, MacLean MR. Effect of tryptophan hydroxylase 1 deficiency on the development of hypoxia-induced pulmonary hypertension. Hypertension. 2007 Jan;49(1):232-6. doi: 10.1161/01.HYP.0000252210.58849.78. Epub 2006 Nov 27. PMID 17130306
- [Result] Sole MJ, Madapallimattam A, Baines AD. An active pathway for serotonin synthesis by renal proximal tubules. Kidney Int. 1986 Mar;29(3):689-94. doi: 10.1038/ki.1986.53. PMID 3702223